CLINICAL TRIAL: NCT01012713
Title: Pilot Open-Label Clinical Trial to Test Efficacy and Safety of Combination of Clobex® Spray With Excimer Laser Therapy [Photomedex XTRAC ® Velocity] in the Treatment of Generalized Plaque Psoriasis Followed by Maintenance With Topical Vectical® Ointment
Brief Title: Safety and Efficacy Study of Combination Treatment With Excimer Laser, Clobex Spray, and Vectical Ointment in the Treatment of Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perfect Storm
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Stable Plaque Psoriasis
Keywords: Psoriasis; Excimer; Laser; Clobex; Vectical; clobetasol spray; calcitriol; Generalized plaque type psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Treatment (Experimental): All patients will receive treatment with Clobex Spray, Vectical Ointment, and Excimer Laser
  Interventions: Drug: Clobex Spray; Drug: Vectical Ointment; Procedure: Excimer Laser

INTERVENTIONS:
Drug: Clobex Spray — Clobex Spray BID for Weeks 1-4 and weeks 9-12
Drug: Vectical Ointment — Vectical ointment BID for weeks 5-8 and 9-12
Procedure: Excimer Laser — Laser treatment for weeks 1-6 study and as needed for patients with less than PASI-75 response thereafter.

SUMMARY:
This is a 12-week, open-label, pilot trial evaluating the efficacy and safety of the combination of Clobex® spray with excimer laser therapy as the initial treatment of generalized plaque psoriasis, followed by maintenance therapy with topical Vectical. The study will be conducted in three distinct periods, namely Period A, Period B, and Period C, each of 4 weeks duration. During Period A (weeks 1 through 4), patients will use Clobex® spray twice daily along with excimer laser treatments twice weekly with the Photomedex XTRAC® Velocity machine. The goal of Period A is to achieve Psoriasis Area Severity Index (PASI) 75 in 100% of patients within four weeks. During Period B (weeks 5 through 8), patients would be treated with topical Vectical® twice daily. Thus, there is a steroid-free interval during which patients will not be using Clobex® spray. The goal of Period B is to maintain the patient's response using only non-steroid options. During Period C of the study, patients will use Clobex® spray BID and Vectical® BID. Period C (weeks 9 through 12) will be a "booster" period in which the goal is to see if 100% of patients can achieve Psoriasis Area Severity Index (PASI) 90-100. Regarding excimer laser therapy: all patients will be receiving excimer laser therapy twice weekly for the first 6 weeks of the study (up to the halfway point) which is 12 excimer laser treatments. At that point, only those patients achieving <Psoriasis Area Severity Index (PASI)75 response will continue to receive twice weekly excimer laser treatments for the remaining 6 weeks of the study.

DETAILED DESCRIPTION:
Psoriasis is an inflammatory skin disease affecting approximately 2% of the population, and approximately one-third of patients experience generalized psoriasis ( ). Current treatment options include topical medications, ultraviolet B and oral psoralen with ultraviolet A phototherapy, biologic agents, non-biologic systemic medications, and combinations of the aforementioned. Phototherapy treatment, although effective for many patients, often is inconvenient, requiring three treatments weekly for 2-3 months in order to achieve significant improvement in a patient's psoriasis. The newer biologic medications, while effective in many patients, work by systemic immunosuppression with increased risk of malignancies, infections including tuberculosis and histoplasmosis, congestive heart failure, lupus-like syndrome, demyelinating diseases, etc. In addition to side effects from systemic immunosuppression, non-biologic systemic agents can have major organ toxicity as a potential side effect including bone marrow suppression, liver toxicity, kidney toxicity, etc.

Currently, we are at the threshold of a new era, where the possibility exists of treating generalized psoriasis with absolute systemic safety and better efficacy than any systemic or biologic agent. This possibility can only become a reality with a "perfect storm," in which three storms collide. This "perfect storm" may achieve a result which no other therapy has yet achieved: a Psoriasis Area Severity Index (PASI)75 response in 100% of patients after only 4 weeks of therapy. The three "storms" include Clobex® spray, Vectical® ointment, and the excimer laser machine XTRAC® Velocity.

Laser therapy (fiberoptically-directed monochromatic UVB light) targets only psoriatic plaques. This allows much more aggressive phototherapy as compared to traditional ultraviolet B and oral psoralen with ultraviolet A , which exposes non-involved skin as well as psoriatic skin to UV light. With aggressive excimer laser therapy, it is well known that psoriasis can improve significantly or clear in approximately ten sessions instead of the 30 to 40 sessions needed with regular full-body phototherapy to achieve clearance of the skin. This dramatic difference is attributed to the fact that psoriatic lesions are able to withstand a much higher dose of light than non-involved skin. Excimer laser therapy dosing is determined by the maximum tolerance of psoriatic skin whereas full body UV therapy dosing is determined by the MED (minimal erythema dose) of non-involved skin. Delivery of higher doses subsequently results in faster clinical response and much greater clinical efficacy. Hence, the new supra-erythemogenic phototherapy strategy results in a fewer number of sessions needed for clearance ( ). The supra-erythemogenic phototherapy strategy involves delivering UVB at a dose much greater than the minimal erythema dose (MED) (2). MED is the traditional limit on how aggressively non-laser phototherapy can be conducted (UVB doses beyond the MED will burn the patient).

In addition, excimer laser therapy results in no photo-damage to non-involved skin, given its targeted application. The Photomedex XTRAC® Velocity is the latest version of the excimer laser, which is 300-400% more powerful than its predecessor, the XTRAC® Ultra machine. This increased power makes treatment of generalized, moderate to severe psoriasis not only feasible but attractive. Time required for each treatment is decreased by one-third, as compared to the XTRAC® Ultra which was previously the most powerful excimer laser machine. XTRAC® Velocity is not yet available: it is scheduled to be introduced in a few months. With XTRAC® Velocity, it is expected that generalized psoriasis patients with 10-30% total body surface involvement can be treated in 10-15 minutes and great improvement can be achieved after approximately just ten laser treatment sessions.

Using the XTRAC® Ultra machine, in a pilot study of 9 patients receiving excimer laser therapy twice weekly for 12 weeks, 77% of patients achieved a Psoriasis Area Severity Index (PASI) 75 response ( ). In another study of 124 patients with stable plaque psoriasis (n = 124) covering less than 10% body surface area (BSA) were enrolled and 80 completed the study ( ). Seventy-two percent of patients achieved at least 75% clearing in an average of 6.2 treatments. Thirty-five percent achieved 90% clearing in an average of 7.5 treatments. In another study of 40 patients treated with the excimer laser under a protocol determined by MED of the involved skin, patients cleared in approximately half the number of treatments compared to patients treated under a protocol where dosage was determined by MED of non-involved skin ( ). However, aggressive laser therapy can also irritate the skin, and Clobex® spray can be an ideal partner to enhance the efficacy and prevent irritation of the skin from aggressive, supra-erythemogenic UVB irradiation. Moreover, beyond prevention of skin irritation, there are additional merits of combining Clobex® spray with excimer laser. These are the following:

* The very real possibility of synergistic efficacy where two very effective, external therapeutic modalities are combined to possibly result in 100% of patients achieving Psoriasis Area Severity Index (PASI) 75 by not week 12, but week 4 of therapy. If this type of efficacy can be demonstrated, it would wipe out all competition in terms of therapeutic efficacy.
* It is tedious to treat multiple small plaques with excimer laser therapy alone. The use of Clobex® ® spray can help eliminate such small psoriatic plaques en masse.
* Laser therapy can help eliminate stubborn plaques still resistant to Clobex® ® spray used BID for one month.

In a study of 1254 subjects treated with clobetasol propionate spray 0.05% as monotherapy twice daily for four weeks, 35.7% of patients achieved clearance and 37.3% of patients were almost clear using a 6-point target plaque severity scale. Additionally, at week 4, 80% of subjects achieved target plaque severity (TPS) success, p<0.001. This was specifically defined as a score of clear, almost clear using the TPS scale or an improvement in severity of 2 grades. Topical steroids have the potential for adrenal suppression. However, when topical steroids are used for one month or less at a time, this transient adrenal suppression that may result is not a clinical problem.Furthermore, when using Clobex® spray, patients are required to have a steroid-free interval after 4 weeks of therapy. The effect of Clobex® spray can be maintained with a safe, non-steroidal topical medication, such as Vectical. This newer Vitamin D topical agent can be used up to 210 g weekly, as compared to topical calcipotriol (Dovonex®) which is limited to 100 g weekly, due to the better safety profile of Vectical. Thus, Vectical can be used for patients with generalized plaque psoriasis covering up to 35% body surface area. In addition, a comparative study in 250 patients demonstrated that Vectical caused significantly less skin irritation as compared to calcipotriol ( ). Thus, with the imminent approval of Vectical, we are entering a new era where a Vitamin D analogue can be used to treat patients with generalized psoriasis. With these three "storms" gathering force, we propose the following study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age of older
2. Subjects should have ≥ 10%, but not more than 20% total body involvement of stable plaque type psoriasis.
3. Subjects must have BMI < 30 and weigh less than 250lbs
4. Subjects must have Fitzpatrick Skin Type II or above (see Attachment A)
5. Subjects must be able to discontinue any topical therapy (other than emollients) or received UVB phototherapy 2 weeks prior to starting the study.
6. Subjects must be able to discontinue any biologic or systemic agents or oral psoralen with ultraviolet A 4 weeks prior to starting the study.
7. Subject is able to complete the study and to comply with study instructions.
8. Subject is capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
9. Any additional diagnoses must, in the investigator's opinion, not preclude the subject from safely participating in this study or interfere with the evaluation of the subject's psoriasis

Exclusion Criteria:

1. Subject is younger than 18 years of age.
2. Subject has less than 10% or greater than 20% body surface involvement of his/her psoriasis.
3. History of known or suspected intolerance to any of the ingredients of the investigational study product.
4. Subject has a photosensitivity disorder (such as lupus, etc.) or a history of clinically significant photosensitivity.
5. Subjects possess other diagnoses that, in the investigator's opinion, preclude him/her from safely participating in this study or interfere with the evaluation of the subject's psoriasis.
6. Subject is not willing to discontinue topical treatment (other than emollients) or UVB phototherapy for 2 weeks prior to starting the study
7. Subject is not willing to discontinue biologic or systemic agents or oral psoralen with ultraviolet A for 4 weeks prior to starting the study.
8. Subject has psoriatic involvement only on the hands, feet, or scalp.
9. Subject has been diagnosed with unstable or non-plaque forms of psoriasis, including guttate, erythrodermic, exfoliative, or pustular psoriasis.
10. Subject has a history of keobnerization phenomenon
11. Subject has keloids or past history of keloid formation
12. Subject has melanoma or past history of melanoma
13. Subject has active (cutaneous) invasive non-melanoma skin cancer (NMSC)
14. Subject is determined not be a candidate for phototherapy by the investigator
15. Subject has used other investigational drugs within 4 weeks prior to the study
16. Subject is known, or suspected of being unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — UCSF Department of Dermatology; Tina Bhutani, MD, Study Director — UCSF Department of Dermatology
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Treatment: All patients will receive treatment with Clobex Spray, Vectical Ointment, and Excimer Laser
  Clobex Spray: Clobex Spray BID for Weeks 1-4 and weeks 9-12
  Vectical Ointment: Vectical ointment BID for weeks 5-8 and 9-12
  Excimer Laser: Laser treatment for weeks 1-6 study and as needed for patients with less than 75% reduction in the Psoriasis Area and Severity Index thereafter.
Period: Overall Study
Arm/Group | Open-Label Treatment
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Groups:
- Open-Label Treatment: All patients will receive treatment with Clobex Spray, Vectical Ointment, and Excimer Laser
  Clobex Spray: Clobex Spray BID for Weeks 1-4 and weeks 9-12
  Vectical Ointment: Vectical ointment BID for weeks 5-8 and 9-12
  Excimer Laser: Laser treatment for weeks 1-6 study and as needed for patients with less than 75% reduction in Psoriasis Area and Severity Index thereafter.
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30
Psoriasis Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index measures the severity of psoriasis on a scale of 0 (no evidence of psoriasis) to 72 (worst possible psoriasis). The score is based on the redness, scaling, thickness and amount of body surface area affected by psoriasis.
  units on a scale | 12.7 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be the Percentage of Patients Achieving a 75% Reduction in the Psoriasis Area and Severity Index at Week 12.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 30
percent | 83 [65 to 94]

2. Secondary Outcome: The Secondary Endpoint Will be the Percentage of Patients Achieving a 75% Reduction in Psoriasis Area and Severity Index at Weeks 4 and 8.
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 30
percent
  Week 8 | 72 [50 to 85]
  Week 4 | 45 [31 to 52]

3. Secondary Outcome: A Tertiary Endpoint Will be the Percentage of Patients Achieving 90% Reduction in Psoriasis Area and Severity Index at Week 12.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Open-Label Treatment: All patients will receive treatment with Clobex Spray, Vectical Ointment, and Excimer Laser
  Clobex Spray: Clobex Spray BID for Weeks 1-4 and weeks 9-12
  Vectical Ointment: Vectical ointment BID for weeks 5-8 and 9-12
  Excimer Laser: Laser treatment for weeks 1-6 study and as needed for patients with less than a 75% reduction in Psoriasis Area and Severity Index.
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 30
percent | 45 [27 to 62]

ADVERSE EVENTS:
Arm/Group | Open-Label Treatment
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment (N=30)
Phototoxicity (Skin and subcutaneous tissue disorders) | 5 (5) — Minor burning, redness or blistering from laser treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No